CLINICAL TRIAL: NCT07159087
Title: A Multicenter, Prospective, Randomized, Double-blind, Pivotal Clinical Trial to Compare the Safety and Efficacy for In-segment Late Lumen Loss of the 'Genoss® SCB' Versus 'SeQuent® Please NEO' in Patients With Coronary ISR
Brief Title: The Safety and Efficacy for In-segment Late Lumen Loss of the 'Genoss® SCB' Versus 'SeQuent® Please NEO' in Patients With Coronary ISR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Genoss Co., Ltd. (Industry)
Collaborators: Synex Consulting Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP-DS2201
Record Dates: First submitted 2025-06-27; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: In-stent Restenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Genoss® SCB (Experimental): Sirolimus Coated PTCA Balloon Catheter
  Interventions: Device: Sirolimus Coated PTCA Balloon Catheter(Genoss® SCB)
- SeQuent® Please NEO (Active Comparator): Paclitaxel Coated PTCA Balloon Catheter
  Interventions: Device: Paclitaxel Coated PTCA Balloon Catheter(SeQuent® Please NEO)

INTERVENTIONS:
Device: Sirolimus Coated PTCA Balloon Catheter(Genoss® SCB) — Drug Coated Balloon
  Arms: Genoss® SCB
Device: Paclitaxel Coated PTCA Balloon Catheter(SeQuent® Please NEO) — Drug Coated Balloon
  Arms: SeQuent® Please NEO

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Genoss® SCB by comparing in-segment late lumen loss (LLL) to the control group (SeQuent® Please NEO) at 6 months in patients with coronary stent-in-stent restenosis (ISR) with a reference vessel diameter of 2.0-4.0 mm.

DETAILED DESCRIPTION:
This pivotal study is a randomized controlled trial to compare with the control group (SeQuent® Please NEO), and will recruit 94 patients with in-stent restenosis (ISR) from 9 institutions. The test group (Genoss® SCB) and the control group (SeQuent® Please NEO) will be randomly assigned 1:1, and all patients will be followed up at 1, 6, and 12 months after the procedure. The primary endpoint is to evaluate in-segment late lumen loss by quantitative coronary angiography (QCA) by an independent assessor at 6 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 19 years of age
* Patients with in-stent restenosis who are candidates for percutaneous coronary intervention (PCI)
* In cases corresponding to one of the following conditions: non-ST-segment elevation myocardial infarction (NSTEMI), stable angina, unstable angina, or silent myocardial ischemia
* Women of childbearing potential* must agree to use at least one medically acceptable method of contraception** throughout the duration of the clinical trial
* Subjects who voluntarily agree to participate and provide written informed consent
* Subjects who are willing to comply with the requirements of the clinical trial protocol
* Subjects who develop in-stent restenosis (ISR) ≥ 90 days after the index coronary stent implantation, with the restenosis classified as Mehran type I to III
* Subjects with a maximum of two ISR lesions, with visually estimated significant coronary artery stenosis on quantitative coronary angiography analysis (QCA) meeting one of the following criteria:

  1. In asymptomatic patients: in-segment percent diameter stenosis (DS%) > 70% compared to the reference vessel diameter of the target vessel* (*Target vessel: the vessel containing the target lesion with the minimum lumen diameter.)
  2. In patients with angina symptoms or evidence of ischemia on non-invasive functional testing: DS% > 50%
* On QCA, the ISR lesion(s) to be treated must have a lesion length < 36 mm and the reference vessel diameter (RVD) of the target coronary artery must be between 2.0 mm and 4.0 mm.

Exclusion Criteria:

* Patients diagnosed with ST-segment elevation myocardial infarction (STEMI) by electrocardiogram.
* Known hypersensitivity or contraindications at screening to any of the following drugs or substances: Aspirin, Heparin, Clopidogrel, Prasugrel, Ticagrelor, Sirolimus, Paclitaxel, Delivery matrix (e.g., shellac, vitamin E-TPGS), Ticlopidine, Contrast agents (e.g., Iopromide) Note: Subjects with contrast media sensitivity may be enrolled if the reaction is manageable with steroids and pheniramine; however, those with a known anaphylactic reaction are excluded.
* Subjects who are scheduled for or require surgery within 1 year of the index procedure that would necessitate discontinuation of antiplatelet therapy.
* Subjects with bleeding disorders, gastrointestinal ulcers, or any conditions that may increase the risk of bleeding, in which anticoagulation is contraindicated or limited.
* Subjects with a left ventricular ejection fraction (LVEF) < 30% as assessed by echocardiography.
* Severe renal failure (Creatinine > 2.0 mg/dL) that makes QCA inappropriate.
* Subjects with cardiogenic shock.
* Pregnant or breastfeeding women: Women of childbearing potential with a positive urine hCG (or serum β-hCG) test are excluded.
* Subjects with an estimated life expectancy of less than 1 year due to comorbid conditions.
* Subjects with medical conditions such as significant psychiatric disorders that may interfere with trial participation or outcomes.
* Subjects who, in the investigator's opinion, are inappropriate for this clinical trial or for whom participation poses increased risk.
* Participation in another clinical trial currently or within 90 days prior to screening.
* Any other condition deemed ethically or clinically inappropriate by the investigator to participate in the study: Specific reasons should be recorded in the Case Report Form (CRF).

[Exclusion Criteria Based on QCA and Pre-Dilatation Assessment of ISR Lesions]

* ISR lesions located in graft vessels following coronary artery bypass grafting (CABG).
* Presence of coronary stent fracture in the ISR lesion to be treated.
* Target lesion with two or more stents implanted, i.e., all segments of the target lesion contain ≥2 layers of stents.
* Presence of additional lesions proximal or clinically significant distal to the target lesion (>2.0 mm RVD) with >50% stenosis.
* Subjects requiring CABG based on any of the following:

  1. Lesions in the left main coronary artery.
  2. Triple-vessel coronary artery disease.
  3. Other conditions requiring CABG as determined by the investigator.
* Subjects for whom pre-dilatation is not feasible or has failed, making application of the investigational device difficult due to any of the following:

  1. Total occlusion of the target lesion.
  2. Evidence of thrombus not treatable with aspiration.
  3. Severe vessel tortuosity or calcification preventing access to the target site, as determined by the investigator.
  4. Other conditions deemed unsuitable for investigational device application by the investigator.
* After lesion pre-dilatation, if any of the following are present:

  1. Need for atherectomy (rotational, orbital, or laser).
  2. Presence of flow-limiting dissection of NHLBI type C or higher requiring stent implantation.
  3. Residual stenosis* in the target lesion. (*Defined as in-segment DS > 30%)
  4. Fractional flow reserve (FFR) ≤ 0.8 (FFR measurement may be omitted at the discretion of the investigator.)
  5. TIMI flow < 3

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
In-segment late lumen loss after procedure | at 6 months after procedure
  In-segment refers to a portion including within 5 mm of each of the distal and proximal portions at the boundary of the inserted stent. Therefore, in-segment late lumen loss (LLL) is defined as the difference (mm) in the minimum lumen diameter (MLD) within the segment at 6 months from baseline.

SECONDARY OUTCOMES:
In-stent late lumen loss after procedure | at 6 months after procedure
  In-stent refers to a portion between each of the distal and proximal portions. Therefore, in-stent late lumen loss (LLL) is defined as the difference (mm) in the minimum lumen diameter (MLD) within the segment at 6 months from baseline. This is assessed by an independent evaluator using quantitative coronary angiography analysis (QCA) imaging.
Target Lesion Failure (TLF), % | at 1 month, 6 months, and 12 months after procedure
  Target lesion failure is defined as a composite of cardiac death, target vessel-related myocardial infarction (TV-MI), and target lesion revascularization (TLR).
Patient-oriented composite endpoint (POCE), % | at 1 month, 6 months, and 12 months after procedure
  POCE is defined as a composite of all-cause death, any myocardial infarction (MI), any revasularization or stroke.
Device success rate, % | Immediately after the procedure
  Device success rate is defined as successful delivery of the device to the target lesion during the procedure, normal inflation, deflation, and catheter withdrawal of the without balloon rupture.
Procedural success rate, % | up to 24 hours
  The definition of procedural success includes the of device success, freedom adverse events in-hospital [cardiovascular death, target lesion revascularization, peri-procedural myocardial infarction, any stroke, and BARC 3-5 bleeding], and freedom from bail-out stenting.
Binary restenosis rate, % | at 6 months after procdure
  defined as a in-segment diameter stenosis ≥ 50% at angiographic follow-up
Cardiac Death, % | at 1 month, 6 months, and 12 months after procedure
  Death caused by acute MI, Sudden cardiac, including unwitnessed, death, Death resulting from heart failure, Death caused by stroke, Death caused by cardiovascular procedures, Death resulting from cardiovascular haemorrhage (haemorrhage deriving from cardiac and/or vascular disease/injuries)
All-cause death, % | at 1 month, 6 months, 12 months after procedure
  Incidence rate of all-cause death including cardiac death.
Target vessel myocardial infarction (TV-MI), % | at 1 month, 6 months, and 12 months after procedure
  Incidence rate of target vessel myocardial infarction
Myocardial infarction (MI), % | at 1 month, 6 months, and 12 months after procedure
  Incidence rate of all myocardial infarction
Ischemia-driven target lesion revascularization (ID-TLR), % | at 1 month, 6 months, and 12 months after procedure
  Target lesion revascularization is defined as a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Ischemia-driven target vessel revascularization (ID-TVR), % | at 1 month, 6 months, and 12 months after procedure
  Target vessel revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel.
Revascularization, % | at 1 month, 6 months, and 12 months after procedure
  Revascularizations are defined according to the vessel/lesion treated and are identified as target or non-target, based on the initial site of the treatment.
Stent thrombosis | at 1 month, 6 months, and 12 months after procedure
  Stent thrombosis will be assessed and classified according to the definitions established by the Academic Research Consortium-2 (ARC-2).
  Stent thrombus is classified based on how the diagnosis is confirmed. These classifications include definite, and probable stent thrombosis.
  Definite stent thrombosis Requires confirmation of stent thrombosis on angiography.
  Probable stent thrombosis Consider if there is active ischemia on electrocardiogram (EKG) or stress in the distribution of prior stent and absence of significant coronary lesion on angiography.
  Timing may be divided between acute, subacute, early, and late.
  When classified as early, or late:
  Early stent thrombosis occurs within one month of initial placement. Late stent thrombosis occurs between 1 and 12 months of initial placement.
  Early stent thrombosis is divided between acute or subacute:
  Acute thrombosis occurs within 24 hours of initial placement. Subacute thrombosis occurs between 24 hours to one month of initial place
Stroke, % | at 1 month, 6 months, and 12 months after procedure
  Neuro-ARC definitions (according to ARC-2 criteria)
Major bleeding BARC type III to V, % | at 1 month, 6 months, and 12 months after procedure
  Major bleeding according to the Bleeding Academic Research Consortium (BARC) scale includes BARC types 3 to 5. Type 3 bleeding encompasses significant bleeding, including overt bleeding with a hemoglobin drop, intracranial hemorrhage, and bleeding requiring surgery or vasoactive agents. Type 4 refers to bleeding related to coronary artery bypass grafting (CABG). Type 5 bleeding is fatal, either probable or definite.
  BARC Type 3: Significant Bleeding 3a: Overt bleeding plus a hemoglobin drop of 3-5 g/dL. 3b: Overt bleeding plus a hemoglobin drop of 3-5 g/dL, cardiac tamponade, surgical intervention required, or intravenous vasoactive agents used.
  3c: Intracranial hemorrhage.
  BARC Type 5: Fatal Bleeding 5a: Probable fatal bleeding, no definitive cause of death but clinically suspected.
  5b: Definite fatal bleeding, confirmed by imaging or autopsy.
Abrupt closure/ Sub abrupt closure, % | at 1 months after procedure
  ① Abrupt closure: Defined as a newly developed, significant reduction in blood flow within the target vessel (TIMI grade 0 or 1) that persists and requires an unplanned rescue strategy (including emergency surgery). This must be associated with mechanical dissection of the treated or manipulated vessel, coronary thrombosis, or severe spasm.
  ② Sub-abrupt closure: Defined as abrupt closure occurring after the index procedure (after the patient has left the procedure room) but before Visit 3 (4 weeks post-procedure).

CONTACTS AND LOCATIONS:
Overall Officials: In-ho Chea, MD, Principal Investigator — Cardiology
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea